CLINICAL TRIAL: NCT01518595
Title: Bosentan for Treatment of Hepatopulmonary Syndrome in Patients With Liver Cirrhosis - a Prospective Double Blind Randomized Controlled Clinical Study
Brief Title: Bosentan for Treatment of Hepatopulmonary Syndrome in Patients With Liver Cirrhosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: too slow patient recruitment
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Valentin Fuhrmann, MD, Associate Professor of Medicine, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-Fuhrmann
Record Dates: First submitted 2011-10-26; First posted 2012-01-26 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Hepatopulmonary Syndrome; Liver Cirrhosis
Keywords: patients
MeSH Terms: conditions — Hepatopulmonary Syndrome; Liver Cirrhosis | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- placebo (Placebo Comparator): Patients will receive placebo tablets twice daily for 3 months.
  Interventions: Drug: Placebo
- bosentan (Active Comparator): pts. will receive bosentan for 3 months
  Interventions: Drug: bosentan

INTERVENTIONS:
Drug: bosentan — pts. will receive bosentan for 3 months
  Arms: bosentan
Drug: Placebo — pts. will receive placebo for 3 months
  Arms: placebo

SUMMARY:
The most common observed cause of gas exchange abnormalities and hypoxemia in cirrhosis is the hepatopulmonary syndrome (HPS) with a reported prevalence of 20-47% in patients with hepatic impairment and cirrhosis. HPS is by far the most frequent respiratory complication of cirrhosis. It is a progressive disease leading to significantly increased mortality. Up to date, the only therapeutic option is liver transplantation. The study hypothesis is that administration of bosentan in patients with liver cirrhosis suffering from hepatopulmonary syndrome improves gas exchange. 18 patients with liver cirrhosis fulfilling criteria of HPS according to the ERS task force criteria will be included in this block randomized, double-blind, placebo controlled study (12 patients will be treated with bosentan, 6 with placebo). Patients will receive bosentan 62,5mg b.i.d. for 4 weeks and 125 mg b.i.d. for 8 weeks or placebo. The duration of the treatment phase of the study is 12 weeks. The primary endpoint is the alteration of gas exchange after 3 months of therapy. The expected duration of the study is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Presence of HPS
* Age ≥ 18 years

Exclusion Criteria:

* Intracardiac shunting
* Pregnancy
* Known hypersensitivity to bosentan
* Use of glyburide
* Use of cyclosporin A
* Elevation of aminotransferase level of > 3 times the upper limit of normal
* Use of rifampicin
* Females of childbearing potential without use of adequate contraception
* Systolic blood pressure < 85 mmHg
* Clinical relevant anemia
* HIV-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
alveolar-arterial oxygen gradient in mmHg | 3 months

SECONDARY OUTCOMES:
presence of HPS | 3 months
  assessment via contrast enhanced transthoracic echocardiography and pulmonary function testing
6 minutes walking distance in m | 3 months
WHO functional class | 3 months
quality of life | 3 months
  we will us the CAT-questionaire for QoL assessment
aminotransferase level (ASAT, ALAT) | 3 months
  Assessment of the aminotransferase levels in U/L
exhanled nitric oxide in parts per billion | 3 months
hepatic venous pressure gradient (HVPG) in mmHg | 3 months
  HVPG will be assessed after inclusion in the study and after 3 months
pulmonary hemodynamics | 3 months
  pulmonary hemodynamics will be assessed after inclusion and after 3 months
mean arterial blood pressue in mmHg | 3 months
partial pressure of arterial oxygen in mmHg | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Valentin H Fuhrmann, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Dpt. of Internal Medicine 3, Div. of Gastroenterology and Hepatology, Vienna, Austria